CLINICAL TRIAL: NCT00358254
Title: Noninvasive Skin Spectroscopy for Diabetes Screening
Status: Completed | Type: Observational
Sponsor: InLight Solutions (Industry)
Collaborators: VeraLight, Inc. (Industry)
Other Study IDs: ILS-04-262
Record Dates: First submitted 2006-07-27; First posted 2006-07-31 (Estimated); Last update posted 2010-07-22 (Estimated); Status verified 2007-11

CONDITIONS: Prediabetic State; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Prediabetic State; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

SUMMARY:
The objective of this study is to assess the performance of a noninvasive device for the early screening of Diabetes Mellitus.

DETAILED DESCRIPTION:
Approximately 18 million people have Type II diabetes, and of these, an estimated thirty-five percent are unaware of their condition. This translates to roughly 6.3 million undiagnosed cases worldwide in 2002. Many diagnoses are made years after the onset of the disease. This allows progression of the vascular lesions that arise during the time of uncontrolled glucose levels. As a result, microvascular retinopathy, nephropathy, and neuropathy are on the rise, as well as macrovascular complications such as: coronary heart disease, and cerebral vascular accidents. The prevalence and trends of diabetes underscore the need for effective and widespread screening. Our fluorescence based system under development will noninvasively measure skin glycation end products that are known to be strongly correlated with diabetes status and complications. Since the test would be painless and require no patient fasting, significant obstacles to screening compliance would be mitigated. The system offers hope for a screening test that is more sensitive and specific than the invasive tests currently used for diabetes screening (Oral Glucose Tolerance Test (OGTT) and the Fasting Plasma Glucose (FPG) test).

ELIGIBILITY:
Inclusion Criteria:

* Volunteers without Diabetes.
* Volunteers at risk for developing Type II diabetes.
* 18 years of age and older.

Exclusion Criteria:

* Under 18 years of age.
* Those diagnosed with Diabetes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Those at risk for diabetes
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2004-10; Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Rohrscheib, M.D., Principal Investigator — UNMHSC
Locations (2):
- United States (2):
  - InLight Solutions, Albuquerque, New Mexico
  - Tricore Reference Laboratory- Presbyterian Professional Building, Albuquerque, New Mexico

REFERENCES:
- See also: Related Info — http://www.inlightsolutions.com
- See also: Related Info — http://www.veralight.com